CLINICAL TRIAL: NCT02392286
Title: A Prospective, Randomized Trial Comparing the Efficacy of Body-weight Based Versus Fixed Corticosteroid Dosage on Remission in Patients With Moderate to Severe Crohn's Disease Flares
Brief Title: Corticosteroid Dosage for Crohn's Disease Flare
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: insufficient enrollment
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1501015143
Record Dates: First submitted 2015-03-12; First posted 2015-03-18 (Estimated); Results first posted 2020-01-22 (Actual); Last update posted 2021-08-09 (Actual); Status verified 2021-08

CONDITIONS: Crohn's Disease; Inflammatory Bowel Disease
Keywords: Corticosteroid
MeSH Terms: conditions — Crohn Disease; Inflammatory Bowel Diseases | interventions — Adrenal Cortex Hormones; Prednisone; Methylprednisolone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Weight-based (Active Comparator): Corticosteroid dose weight-based at equivalent to 1mg/kg prednisone daily.
  Interventions: Drug: Corticosteroid
- Fixed dose (Active Comparator): Corticosteroid dose fixed at equivalent to 40mg prednisone daily.
  Interventions: Drug: Corticosteroid

INTERVENTIONS:
Drug: Corticosteroid — Subjects will receive prednisone orally; if intravenous corticosteroid required initially they will receive methylprednisolone for the first 3-4 days of therapy.
  Other Names: Prednisone; Methylprednisolone

SUMMARY:
Prospective randomized comparative effectiveness trial designed to compare fixed dosing and weight-based dosing of corticosteroids in patients with Crohn's disease flares.

DETAILED DESCRIPTION:
* Determine if weight-based corticosteroid (1mg/kg daily) induces remission at a greater rate than fixed corticosteroid dosage.
* Determine if weight-based corticosteroid is associated with greater rate of adverse events than fixed corticosteroid dosage.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18
* Established diagnosis of Crohn's disease
* Diagnosis of Crohn's flare
* Decision by treating gastroenterologist to start corticosteroid therapy

Exclusion Criteria:

* Patients in whom corticosteroid therapy is contraindicated: immunocompromised (active cancer on chemotherapy or radiation treatment), severe liver disease (decompensated cirrhosis, active alcoholic hepatitis), end-stage renal disease on dialysis, AIDS or AIDS-defining illness; myocardial infarction within the past year; NYHA Class 4 heart failure
* Patients on systemic corticosteroid therapy currently or within the past 8 weeks
* Patients not on stable doses of immunomodulators or biologics for at least 8 weeks
* Infectious colitis (e.g., C. difficile, CMV, HSV)
* Systemic infections (bacteremia, fungal infections)
* Fulminant Crohn's disease
* Patients who require imminent surgery
* Abscess
* Pregnancy
* Weight <35 kg

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2015-03 (Actual); Primary Completion 2016-12-19 (Actual); Study Completion 2016-12-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Loren Laine, MD, Principal Investigator — Yale University, Section of Digestive Diseases
Locations (1):
- Yale-New Haven Hospital, New Haven, Connecticut, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Weight-based | Fixed Dose
Started | 7 | 8
Completed | 4 | 6
Not Completed | 3 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Weight-based | Fixed Dose | Total
Number analyzed (Participants) | 7 | 8 | 15
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 5 | 6 | 11
  >=65 years | 2 | 2 | 4
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 4 | 7
  Male | 4 | 4 | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 6 | 8 | 14
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 7 | 7 | 14
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 7 | 8 | 15

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants in Remission at End of 2 Weeks
Description: Number of participants with Harvey Bradshaw Index < 5 at end of 2 weeks. The minimum score obtainable is 0, suggesting absence of disease or remission, while the maximum score obtainable goes beyond 18 points, depending on the number of stools the patient identifies per day (because 1 point is given for each stool in a day, there is no specific maximum score. A higher score represents more severe disease. <5 is determined to be remission.
Time Frame: 2 weeks
Population: 1 patient in fixed dose group did not return for this assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | Weight-based | Fixed Dose
Number analyzed (Participants) | 7 | 7
Participants | 2 | 3

2. Secondary Outcome: Number of Participants With Response at End of 2 Weeks
Description: Number of participants with at least a 3-point drop in Harvey-Bradshaw Index at end of 2 weeks
Time Frame: 2 weeks
Population: 1 patient in fixed-dose group did not return for this assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | Weight-based | Fixed Dose
Number analyzed (Participants) | 7 | 7
Participants | 4 | 6

3. Secondary Outcome: Number of Participants With Response or Remission at End of 1 Week
Description: Number of participants with Harvey-Bradshaw Index <5 or with a drop in Harvey-Bradshaw Index of at least 3 points at end of 1 week
Time Frame: 1 week
Population: 1 patient in weight-based group and 2 patients in fixed-dose group did not return for this assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | Weight-based | Fixed Dose
Number analyzed (Participants) | 6 | 6
Participants | 5 | 5

4. Secondary Outcome: Number of Participants With Response or Remission at End of 4 Weeks
Description: Number of participants with Harvey-Bradshaw Index <5 or with a drop in Harvey-Bradshaw Index of at least 3 points at end of 4 weeks
Time Frame: 4 weeks
Population: 2 patients in weight-based group and 1 patient in fixed-dose group did not return for this assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | Weight-based | Fixed Dose
Number analyzed (Participants) | 5 | 7
Participants | 5 | 5

5. Secondary Outcome: Number of Participants With Response or Remission at End of 12 Weeks
Description: Number of participants with Harvey-Bradshaw Index <5 or with a drop in Harvey-Bradshaw Index of at least 3 points at end of 12 weeks
Time Frame: 12 weeks
Population: 1 patient in fixed-dose group did not return for this assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | Weight-based | Fixed Dose
Number analyzed (Participants) | 7 | 7
Participants | 5 | 7

6. Secondary Outcome: Number of Participants With Corticosteroid-associated Side Effects
Description: Number of participants with side effects that may be associated with use of corticosteroids such as mood swings, sleep disturbance, edema, acne, bruising, myalgias.
Time Frame: 12 weeks
Population: 1 patient in fixed dose did not return and did not have any assessment for this outcome after randomization.
Measure: Count of Participants; unit: Participants
Arm/Group | Weight-based | Fixed Dose
Number analyzed (Participants) | 7 | 7
Participants | 5 | 7

ADVERSE EVENTS:
Time Frame: Up to 12 weeks.
Arm/Group | Weight-based | Fixed Dose
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/8
Serious Adverse Events (participants affected / at risk) | 1/7 | 4/8
Other Adverse Events (participants affected / at risk) | 5/7 | 7/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Weight-based (N=7) | Fixed Dose (N=8)
Hospitalization for Crohn's disease (Gastrointestinal disorders) | 1 | 4
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Weight-based (N=7) | Fixed Dose (N=8)
Mood swings (Psychiatric disorders) | 2 | 5
Sleep disturbance (Psychiatric disorders) | 4 | 3
Edema (Endocrine disorders) | 1 | 3
Acne (Skin and subcutaneous tissue disorders) | 2 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 3 | 1
Bruising (Skin and subcutaneous tissue disorders) | 1 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes